CLINICAL TRIAL: NCT00798187
Title: Efficacy of Cancer Support Programs: A Social Comparison Theory Analysis
Status: Terminated | Type: Observational
Why Stopped: Terminated at time of CR - 3.26.2019 - JA
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0594; 1R21CA126854 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Breast Cancer; Behavioral Intervention; Cancer Support Programs; Social Comparison; Heterogeneous support group; Homogeneous support group
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Homogeneous Support Group
  Interventions: Behavioral: Group Meetings; Behavioral: Questionnaire
- Heterogeneous Support Group One
  Interventions: Behavioral: Group Meetings; Behavioral: Questionnaire
- Heterogeneous Support Group Two
  Interventions: Behavioral: Group Meetings; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Group Meetings — 10 weekly group meetings lasting 2 hours.
Behavioral: Questionnaire — Surveys

SUMMARY:
The goal of this research study is to learn if a support group program is acceptable for patients with prostate cancer or patients with breast cancer. Researchers also want to learn if the characteristics of the members of the support group program can have an effect on the quality of life of other members of the support group program. Support group programs will be conducted separately for prostate cancer patients and breast cancer patients.

DETAILED DESCRIPTION:
Screening Questionnaires:

Signing this consent form does not mean that you will be able to take part in this study. You will complete some questions about your mood to help researchers decide if you are eligible to take part in this study. It will take 10 to 15 minutes to complete these questions.

The researcher will discuss the questionnaire results with you and provide you with a list of community referrals and resources.

If your responses to the questions show that you are distressed, you will be eligible to take part in this study. If your responses to the questions show that you are not distressed, you will be randomly selected (as in the flip of a coin) to take part in this study.

If your responses to the questions show that you may harm yourself, a licensed psychologist will follow-up with you and make recommendations for future treatment.

Study Questionnaires:

If you are found to be eligible and are selected to take part in this study, you will be asked to complete questionnaires that will have questions about your medical history, quality of life, mood, thought processes, methods of coping with the disease, and support that you receive from others. It will take about 1 hour to complete these questionnaires.

Support Groups:

You will also take part in a support group program for either prostate or breast cancer patients. Each support group will be made up of about 10 members. Each group will meet 1 time each week for 10 weeks. Each meeting will last about 2 hours. At each meeting, patients will discuss and learn about methods of coping with the disease and ways to relax.

All meetings will be audio-recorded. Recordings will be reviewed by the research team to make sure that the groups are covering the program content.

Length of Study:

You will be on study for about 3 months.

End-of Study Questionnaires:

After the last support group meeting, you will complete questionnaires that will ask questions about your medical history, quality of life, mood, thought processes, methods of coping with the disease, and support that you receive from others. You will be off study after you have completed the end-of-study questionnaires.

This is an investigational study.

Up to 240 patients will take part in this study. Up to 204 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of prostate or breast cancer, regardless of treatment
2. No evidence of metastatic disease
3. Able to read, speak, and write English
4. Resides within one hour of M.D. Anderson Cancer Center
5. 21 years of age or older
6. Able to provide meaningful informed consent as judged by a research team member
7. Being a distressed patient: a T score greater than or equal to 63 on the Global Severity Index (GSI) of the Brief Symptom Inventory (BSI) or a T score greater than or equal to 63 on any two primary dimensions of this measure, or being a non-distressed patient: a T score of < 63 on the GSI and a T score of <63 on all primary dimensions of the BSI.

Exclusion Criteria:

1) None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants, 21 years of age or older, diagnosed with Prostate Cancer or Breast Cancer.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Patient Psychological Functioning and Quality of Life (QOL) | Baseline and Month 3: Questionnaires & Support Group Assessments

SECONDARY OUTCOMES:
To study if the characteristics of the members of the support group program can have an effect on the quality of life of other members of the support group program. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Carmack Taylor, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org